CLINICAL TRIAL: NCT00560495
Title: The Combination of Radiotherapy With the Anti-Angiogenic Agent Tetrathiomolybdate (TM) in the Treatment of Stage I-IIIB Non-Small Cell Lung Cancer (NSCLC): A Phase I Study
Brief Title: Radiation Therapy and Ammonium Tetrathiomolybdate in Treating Patients With Stage I, Stage II, or Stage III Non-Small Cell Lung Cancer
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000574135; RPCI-EPR-38104
Record Dates: First submitted 2007-11-16; First posted 2007-11-19 (Estimated); Last update posted 2022-10-03 (Actual); Status verified 2022-09

CONDITIONS: Lung Cancer
Keywords: stage I non-small cell lung cancer; stage II non-small cell lung cancer; stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer; adenocarcinoma of the lung; adenosquamous cell lung cancer; large cell lung cancer; squamous cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Adenocarcinoma of Lung | interventions — tetrathiomolybdate; Immunoenzyme Techniques; Technetium Tc 99m Sestamibi; Radiotherapy

INTERVENTIONS:
Drug: ammonium tetrathiomolybdate — 4 times daily for up to 3 weeks
Other: immunoenzyme technique
Other: laboratory biomarker analysis
Radiation: Tc 99m sestamibi
Radiation: radiation therapy — once daily, 5 days a week, for 6-7 weeks

SUMMARY:
RATIONALE: Ammonium tetrathiomolybdate may stop the growth of non-small cell lung cancer by blocking blood flow to the tumor. Radiation therapy uses high-energy x-rays to kill tumor cells. Giving ammonium tetrathiomolybdate together with radiation therapy may kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects of giving radiation therapy together with ammonium tetrathiomolybdate in treating patients with stage I, stage II, or stage III non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To assess the acute toxicity of combining antiangiogenic copper reduction with ammonium tetrathiomolybdate (TM) and standard external-beam radiotherapy in patients with stage I-IIIB non-small cell lung cancer.

Secondary

* To measure changes in biological markers of angiogenesis (i.e., ELISA analysis of serum bFGF, VEGF, TGF-beta, IL-6, and IL-8) affected by TM or radiotherapy and an imaging technique (technetium 99m sestamibi) known to correlate with intratumoral angiogenesis.
* To follow the late toxicity that exists when angiogenic inhibition with the copper reduction agent TM is combined with standard external-beam radiotherapy in these patients.
* To collect tumor response, recurrence rate, and survival data on these patients.

OUTLINE:

* Induction phase: Patients receive oral ammonium tetrathiomolybdate (TM) 4 times daily for up to 3 weeks.
* Radiotherapy: Patients undergo radiotherapy once daily, 5 days a week, for 6-7 weeks along with concurrent TM.
* Maintenance phase: Patients continue to receive TM for a total of 1 year . Blood is collected periodically for analysis of laboratory outcomes by ELISA and technetium 99m sestamibi scans. Biomarkers may include VEGF, bFGF, TGF-beta, interleukin (IL)-6, and IL-8.

After completion of study therapy, patients are followed every 3 months for up to 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed non-small cell lung cancer (NSCLC) meeting the following criteria:

  * Squamous, large cell undifferentiated, or adenocarcinoma

    * Sputum cytology not acceptable evidence of cell type
    * Cytologic specimens obtained by brushing, washing, or needle aspiration of a defined lesion allowed
  * Stage I-IIIB disease
  * No evidence of distant metastases
* Planning to receive definitive radiotherapy alone or post-operative radiotherapy (for gross residual disease or positive margin)
* Medically inoperable disease or chemotherapy or surgery refused
* Mediastinal lymph nodes must be evaluated by either mediastinoscopy or by PET scan, unless definitive CT-positive mediastinal disease is noted

  * If patient cannot tolerate mediastinoscopy and no PET is available, the technetium 99m sestamibi scan is allowed for assessment of the mediastinum
* No stage IIIB disease with pleural effusions or stage IV disease
* No small cell lung cancer or mixed small cell/non-small cell histology

PATIENT CHARACTERISTICS:

* SWOG performance status 0-2
* Hemoglobin ≥ 9.0 g/dL
* WBC ≥ 3,000/mm³
* ANC ≥ 1,200/mm³
* Platelet count ≥ 80,000/mm³
* Creatinine < 1.8 mg/dL
* Prior malignancy allowed if disease free for ≥ 5 years

  * Nonmelanoma skin cancer allowed within 5 years
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No grade 3 hemoptysis (or hemoptysis not requiring transfusion, but where the radiation oncologist has concerns about a 3-week delay in treatment)
* No pneumonia due to bronchial obstruction (or a high-grade bronchial obstruction where the radiation oncologist has concerns about a 3-week delay in treatment)
* No transfusion dependence requiring > 2 units of packed RBCs every 2 weeks for more than 28 days
* No medically serious acute or chronic medical condition that is unstable and/or requires intensive management

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Prior thoracic radiation allowed if the new lesion can be treated with absolutely no overlap of previous treatment fields
* At least 3 weeks since prior surgery
* No concurrent chemotherapy

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-05; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Acute toxicity

SECONDARY OUTCOMES:
Assessment of markers of angiogenesis in serum (VEGF, bFGF, TGF-beta, IL-6, IL-8)
Assessment of markers of angiogenesis on imaging (technetium 99m sestamibi) scans
Late toxicity
Collection of response, recurrence, and survival data | every 3 months for up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad K. Khan, MD, PhD, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States